CLINICAL TRIAL: NCT02485444
Title: Oxytocin Infusion vs. Spontaneous Follow-up for Third-stage Management After Second-trimester Abortion: A Randomized Clinical Trial
Brief Title: Oxytocin Infusion vs. Spontaneous Follow-up for Third-stage of Labor After Second-trimester Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-80
Record Dates: First submitted 2015-06-28; First posted 2015-06-30 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Abortion, Induced; Labor Stage, Third/Drug Effects; Pregnancy Trimester, Second; Oxytocin/Administration & Dosage
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin
- Observation (No Intervention)

INTERVENTIONS:
Drug: Oxytocin — 20 IU oxytocin in 500 ml normal saline will be infused 100 ml/h i.v. after fetus is delivered
  Other Names: Synpitan; Pitocin
  Arms: Oxytocin

SUMMARY:
This study compares oxytocin infusion to spontaneous follow-up for third-stage of labor at induced mid-trimester abortions. Patients will be randomized to oxytocin infusion or observation with no pharmacologic intervention. Primary outcome of the study is complete abortion rate within two hours of fetal delivery.

ELIGIBILITY:
Inclusion Criteria:

-Women who had mid-trimester termination of pregnancy between 13-24 gestational weeks

Exclusion Criteria:

* If fetus and placenta expelled together
* Obstetrical haemorrhage needs intervention
* Known prostaglandin allergy

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Complete abortion rate | within 5 minute after placenta delivered
  expulsion of placenta completely without an instrumental assistance within two hours after delivery of fetus

SECONDARY OUTCOMES:
Blood loss estimated by gravimetric method | within 10 minutes after delivery of placenta
  blood loss will be estimated by gravimetric method
Transfusion rate | Within 7 days of hospitalization
  number of packed red cell units transfused
Change in hemoglobin measured by difference in hemoglobin before and 24-hour after abortion | 24 hours after delivery of placenta
  Difference in hemoglobin before and 24-hour after abortion
Placenta delivery time measured by time elapsed until the delivery of the placenta from the delivery of foetus | 5 minute after delivery of placenta
  The time elapsed until the delivery of the placenta from the delivery of foetus

CONTACTS AND LOCATIONS:
Overall Officials: Omer E Yapca, MD, Study Chair — Ataturk University; Ragıp A AL, MD, Principal Investigator — Ataturk University
Locations (1):
- Atatürk Üniversitesi Araştırma Hastanesi, Erzurum, Turkey (Türkiye)